CLINICAL TRIAL: NCT04698330
Title: Effects of Berberine Plus Inulin on Diabetes Care in Patients With Latent Autoimmune Diabetes in Adults: A Randomized Controlled Trial
Brief Title: Effects Of Berberine Plus Inulin On Diabetes Care in Patients With LADA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Yang Xiao, Associate Professor, Department of Metabolism and Endocrinology, Institute of Metabolism and Endocrinology, National Clinical Research Center for Metabolic Diseases, Second Xiangya Hospital, Central South University, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020LADACP
Record Dates: First submitted 2021-01-02; First posted 2021-01-06 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Type 1 Diabetes Mellitus; Autoimmune Diabetes
Keywords: LADA; Berberine; Inulin; Diabetes Care
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Berberine; Inulin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): LADA patients are assigned to receive berberine and inulin for 3-month.
  Interventions: Drug: Berberine; Drug: Inulin
- Group B (Experimental): LADA patients are assigned to receive berberine and placebo(for inulin) for 3-month.
  Interventions: Drug: Berberine; Drug: Inulin placebo tablets
- Group C (Experimental): LADA patients are assigned to receive placebo(for berberine) and inulin for 3-month.
  Interventions: Drug: Inulin; Drug: Berberine placebo tablets
- Group D (Placebo Comparator): LADA patients are assigned to receive placebo(for berberine) and placebo(for inulin) for 3-month.
  Interventions: Drug: Berberine placebo tablets; Drug: Inulin placebo tablets

INTERVENTIONS:
Drug: Berberine — 0.6g (6 pills) of Berberine tablets administered twice a day orally before meal for 3 months
  Arms: Group A; Group B
Drug: Inulin — 0.6g (6 pills) of Inulin tablets administered twice a day orally before meal for 3 months
  Arms: Group A; Group C
Drug: Berberine placebo tablets — 0.6g (6 pills) of Berberine placebo tablets administered twice a day orally before meal for 3 months
  Arms: Group C; Group D
Drug: Inulin placebo tablets — 0.6g (6 pills) of Inulin placebo tablets administered twice a day orally before meal for 3 months
  Arms: Group B; Group D

SUMMARY:
The primary purpose of this study is to evaluate the effects of oral berberine (BBR) and inulin combined with insulin therapy on diabetes care in patients with LADA.

DETAILED DESCRIPTION:
Latent autoimmune diabetes in adults (LADA) is a hybrid form of diabetes, characterized by autoimmune destruction of pancreatic β-cells as well as insulin resistance and is triggered by environmental factors in the context of genetic susceptibility. Meanwhile，blood glucose management is the cornerstone of diabetes care and poor glycemic control will cause a series of diabetes complications. This study will focus on improving the quality of life of LADA patients and blood glucose management as the starting point to explore the improvement effects of combined drugs on the development of diabetes.

Inulin is a common prebiotic that has been shown to improve glycemic control, alter the gut microbiota and suppress inflammation. Berberine(BBR), a small alkaloid isolated from medicinal plants, has been reported to have many therapeutic effects, including anti-bacteria, anti-diabetes, and lipid-lowering. Besides, studies revealed that BBR exerts antidiabetic effects by modulating gut microbiota. In a multicentre, randomized, double-blinded, placebo-controlled 12-week clinical trial conducted in 409 drug-naive T2D patients, Wang et al. confirmed the hypoglycaemic effect of BBR in Chinese participants and demonstrated the BBR-induced changes in the human gut microbiome in comparison with the placebo. Moreover, Ho et al. conducted a randomized, placebo-controlled trial in 38 children with type 1 diabetes using placebo or prebiotic oligofructose-enriched inulin for 12 weeks, and found that oral supplement of the prebiotic could improve glycemic status and β cell function. So we speculate that BBR and inulin combination can also improve glycemic control in the patients with LADA.

This study is a prospective, randomized, double-blind, placebo-controlled trial. The study comprises once screening, the 1-month run-in period, the 3-month treatment period and the 9-month follow-up period. After obtaining the informed consent from the patient who is willing to participate the 3-month treatment will enter to the 1-month run-in period. According to the inclusion/exclusion criteria, the eligible patients will be randomized to the 3-month treatment period. Patients will be randomized into four groups : BBR-alone, inulin+BBR, inulin-alone, or placebo. The primary outcome is to assess the change in glycated hemoglobin levels. Dynamic blood glucose parameters, β-cell function and gut microbiota, as well as adverse events and quality of life will be monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes diagnosed according to the report of WHO in 1999；
2. Meet the Chinese Diabetes Society diagnostic criteria (2012) for LADA: (1)glutamic acid decarboxylase antibody (GADA) positive; (2) age at diagnosis ≧ 18 years old; (3) independent on insulin for more than 6 months after diagnosis;
3. Aged between 18 and 70 years old;
4. 7.0%≤HbA1c ≤10.0%;
5. BMI ≥ 18.5 kg/m2, and no more than 37.5 kg/m2;
6. Written informed consent from the patient or family representative.

Exclusion Criteria:

1. Severe liver dysfunction (ALT and AST greater than 3 times the upper limit of detection);
2. eGFR < 50ml/(min • 1.73 m2);
3. Evidence of acute or chronic infection affecting glycemic control within 4 weeks prior to the first visit;
4. History of any malignancy;
5. Pregnancy, breastfeeding, or planned pregnancy during the study period;
6. Secondary diabetes;
7. Presence of acute complications (ketoacidosis, lactic acidosis or hyperosmolar coma);
8. Severe organic heart disease, including but not limited to congenital heart disease, rheumatic heart disease, hypertrophic or dilated cardiomyopathy, etc., New York Heart Association (NYHA) heart function classification ≥Grade III;
9. Chronic use of systemic glucocorticoids or other immunosuppressive agents for over 3 months，or use of antibiotic medications or other interventions that could affect the gastrointestinal tract for 2 months before the screening and during the whole study period.
10. History of hemolytic anemia or glucose-6-phosphate dehydrogenase deficiency.
11. Allergic to berberine or any components in the combinations.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | 1 year after start of trial
  The primary outcome measure is the change in mean HbA1c level, reflecting the blood glucose management status of the patients.

SECONDARY OUTCOMES:
Change in C-peptide | 1 year after start of trial
  C-peptide are measured before and after a mixed meal tolerance test.
Incidence of acute and chronic diabetes complications | 1 year after start of trial
  In this study, the chronic diabetes complications recorded mainly include diabetic macrovascular disease, diabetic nephropathy, diabetic retinopathy and peripheral neuropathy.
Change in gut permeability | 1 year after start of trial
  Gut permeability is measured by amount of mannitol and lactulose in urine.
Change in gut microbiota composition | 1 year after start of trial
  The changes of gut microbiota are mainly detected by multi omics technology.
Assessment of quality of life | 1 year after start of trial
  Quality of life will be assessed by the Chinese version of the Audit of Diabetes Dependent Quality of Life (ADDQoL-19).
Gastrointestinal side effects and other drug-related side effects | 1 year after start of trial
  The gastrointestinal side effects need to be self-reported by the patient, such as nausea, vomiting, diarrhea, constipation, flatulence, etc.
Hypoglycemic events | 1 year after start of trial
  Hypoglycemia events are divided into mild hypoglycemia and severe hypoglycemia.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Xiao, MD/PhD, Principal Investigator — Institute of Metabolism and Endocrinology, Second Xiangya Hospital, Central South University, China
Locations (1):
- Institute of Metabolism and Endocrinology, Second Xiangya Hospital, Central South University, Changsha, Hunan, China

REFERENCES:
- [Background] Zhang Y, Gu Y, Ren H, Wang S, Zhong H, Zhao X, Ma J, Gu X, Xue Y, Huang S, Yang J, Chen L, Chen G, Qu S, Liang J, Qin L, Huang Q, Peng Y, Li Q, Wang X, Kong P, Hou G, Gao M, Shi Z, Li X, Qiu Y, Zou Y, Yang H, Wang J, Xu G, Lai S, Li J, Ning G, Wang W. Gut microbiome-related effects of berberine and probiotics on type 2 diabetes (the PREMOTE study). Nat Commun. 2020 Oct 6;11(1):5015. doi: 10.1038/s41467-020-18414-8. PMID 33024120
- [Background] Ho J, Nicolucci AC, Virtanen H, Schick A, Meddings J, Reimer RA, Huang C. Effect of Prebiotic on Microbiota, Intestinal Permeability, and Glycemic Control in Children With Type 1 Diabetes. J Clin Endocrinol Metab. 2019 Oct 1;104(10):4427-4440. doi: 10.1210/jc.2019-00481. PMID 31188437
- [Derived] Zhang R, Xiao Y, Yan J, Yang W, Wu X, Mei Z, Zhou Z. Effects of Berberine Plus Inulin on Diabetes Care in Patients With Latent Autoimmune Diabetes in Adults: Protocol for a Randomized Controlled Trial. Front Endocrinol (Lausanne). 2022 Jun 15;13:876657. doi: 10.3389/fendo.2022.876657. eCollection 2022. PMID 35784546